CLINICAL TRIAL: NCT03686072
Title: Head of Glaucoma, Clinical Professor
Brief Title: Cataract Surgery Combined With Endoscopic Goniosynechialysis for Advanced Primary Angle Closure Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Department of Catract, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QZB-HZ-PHACO-EGSL
Record Dates: First submitted 2018-09-21; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Glaucoma, Closed-Angle
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Cataract Extraction

ARMS (1):
- Cataract surgery with goniosynechialysis (Other)
  Interventions: Procedure: Cataract surgery with endoscopic goniosynechialysis

INTERVENTIONS:
Procedure: Cataract surgery with endoscopic goniosynechialysis — Phacoemulsification was performed first. Immediately after implantation of the IOL, a 23G ophthalmic endoscope (OE) probe was inserted into the anterior chamber to visualize the PAS through the main incision and side incision. A viscoelastic agent and a blunt iris spatula were used to release the areas where where PAS existed.

SUMMARY:
In this prospective study, consecutive patients with advanced PACG and cataract who underwent Phaco-IOL-EGSL were invited to participate.

Inclusion and exclusion criteria Inclusion criteria included: a diagnosis of PACG according to the International Society of Geographical & Epidemiological Ophthalmology (ISGEO) diagnostic criteria,14 visual field score ≥18 calculated (as per the method used in the Advanced Glaucoma Intervention Study [AGIS]),15 treatment with IOP-lowering drugs for more than 3 months, and mild to moderate cataract. Exclusion criteria included: secondary angle-closure glaucoma and previous history of surgery, except laser peripheral iridotomy.

Preoperative and postoperative examinations Preoperative examinations included: best corrected logMAR visual acuity (BCVA), number of intraocular pressure (IOP) lowering drugs, slit lamp and fundus examination, gonioscopy, Goldmann applanation tonometry and ultrasound biomicroscopy (UBM). Visual field tests were conducted with a Humphrey Visual Field Analyzer II.

All patients were reviewed at 1 week, 1 month, 3 months, 6 months and 12 months after surgery. The number of IOP-lowering drugs and IOP was observed and recorded at each follow-up. The extent of peripheral anterior synechiae , the BCVA and the visual field were recorded at 12 months following surgery.

Surgery procedure All patients used IOP-lowering drugs before surgery; IOP was controlled under 21mmHg where possible. If the preoperative IOP was over 40mmHg a preoperative anterior chamber paracentesis was performed. All surgeries were performed by the same experienced surgeon (WP). Intraoperative and postoperative complications were recorded.

In all patients, phacoemulsification was performed first. After implantation of the IOL, an ophthalmic endoscope (OE) probe was inserted into the anterior chamber to visualize the PAS through the main incision and side incision. A viscoelastic agent was injected towards the root of the iris where PAS existed. Then a blunt iris spatula was used to release the areas where PAS remained under direct view with the OE. Complete synechialysis was confirmed under the direct view with the OE at the end of the procedure.

Success criteria Based on the AGIS study, we defined surgical success as follows: (1) Standard A: IOP<14mmHg using none or one type of IOP-lowering drug; (2) Standard B: IOP <18mmHg using none or one type of IOP-lowering drug.

DETAILED DESCRIPTION:
Introduction The prevalence of primary angle-closure glaucoma (PACG) is approximately 0.1% of the general population over 40 years of age but up to 1.5% of the Chinese population over 50 years of age. Studies predict that the number of cases of PACG in Asia will increase by 2040.4 Because PACG appears to cause blindness more frequently than primary open-angle glaucoma (POAG), it is considered to be the main cause of binocular glaucoma blindness and reduced quality of life in China. Early diagnosis of PACG is difficult; advanced cases at presentation are not uncommon.

In recent years cataract surgery (phacoemulsification with intraocular lens implantation) combined with goniosynechialysis (Phaco-IOL-GSL) has become more widely used in the treatment of PACG.8-11 Compared with the classic glaucoma filtration surgery, Phaco-IOL-GSL does not involve the creation of a filtering bleb with the need for long-term close follow-up. This is important for patients with poor compliance or difficulty with travel. However, the efficacy and risk of Phaco-IOL-GSL in patients with advanced glaucoma has not been reported. We prospectively performed phacoemulsification combined with intraocular lens implantation combined with endoscopic goniosynechialysis (Phaco-IOL-EGSL) in patients with advanced angle-closure glaucoma, and explored the efficacy and risk of the surgery.

Materials and methods Subjects Our objective was to measure the extent of PAS, number of intraocular pressure(IOP) lowering drugs, IOP, BCVA and visual field before and after surgery in patients with advanced PACG, to investigate the efficacy and safety of Phaco-IOL-EGSL. We also evaluate the correlation between the two groups of data.

In this prospective study, consecutive patients with advanced PACG and cataract who underwent Phaco-IOL-EGSL were invited to participate. The study was approved by the Ethics Committee of the Affiliated Eye Hospital of Wenzhou Medical University and informed consent was obtained from all patients, adhered to the tenets of the Declaration of Helsinki. All patients were treated at the Affiliated Eye Hospital of Wenzhou Medical University between February 2014 and March 2016. A total of 17 subjects (19 eyes) were enrolled in the study. Patients were followed up for 12 months. One patient was lost during follow-up, and 16 subjects (18 eyes) were analyzed in this study. No patient refused to participate in the study.

Inclusion and exclusion criteria Inclusion criteria included: a diagnosis of PACG according to the International Society of Geographical & Epidemiological Ophthalmology (ISGEO) diagnostic criteria,14 visual field score ≥18 calculated (as per the method used in the Advanced Glaucoma Intervention Study [AGIS]), treatment with IOP-lowering drugs for more than 3 months, and mild to moderate cataract. Exclusion criteria included: secondary angle-closure glaucoma and previous history of surgery, except laser peripheral iridotomy.

Preoperative and postoperative examinations Preoperative examinations included: best corrected logMAR visual acuity (BCVA), number of intraocular pressure (IOP) lowering drugs, slit lamp and fundus examination, gonioscopy, Goldmann applanation tonometry and ultrasound biomicroscopy (UBM) (Suowei, Tianjin, China). Visual field tests were conducted with a Humphrey Visual Field Analyzer II (central 30-2 threshold test, size III white stimulus, and SITA-FAST strategy, with the foveal threshold test turned on).

Gonioscopy was performed in a dark room by the same experienced glaucoma specialist (WP) using a Zeiss-style 4-mirror lens (Zeiss Corp, Germany). The examination start with the inferior angle by looking through the superior mirror, the corneal wedge is used to orient oneself to the anatomy.16 The extent of PAS was evaluated by performing indentation gonioscopy around the entire circumference of angle.

All patients were reviewed at 1 week, 1 month, 3 months, 6 months and 12 months after surgery. The number of IOP-lowering drugs and IOP was observed and recorded at each follow-up. The extent of peripheral anterior synechiae , the BCVA and the visual field were recorded at 12 months following surgery.

Surgery procedure All patients used IOP-lowering drugs before surgery; IOP was controlled under 21mmHg where possible. If the preoperative IOP was over 40mmHg a preoperative anterior chamber paracentesis was performed. All surgeries were performed by the same experienced surgeon (WP). Intraoperative and postoperative complications were recorded.

Anaesthesia consisted of topical 0.5% proparacaine and a peribulbar block with bupivacaine. Then conventional phacoemulsification and IOL implantation (CT ASPHINA 509M, Zeiss Corp.) were performed. In all patients, phacoemulsification was performed using the following fluidic parameters: bottle height between 70 and 90 cm, a fixed aspiration flow rate (AFR) of 20 cc/min, and vacuum settings up to 350 mmHg, depending on the grade of nuclear sclerosis. Immediately after implantation of the IOL, a 23G ophthalmic endoscope (OE) probe (URAM E2, USA ENDO OPTIKS) was inserted into the anterior chamber to visualize the PAS through the main incision and side incision. A viscoelastic agent was injected towards the root of the iris where PAS existed (Figure 1A). Then a blunt iris spatula was used to release the areas where PAS remained. The tip was gently moved anteroposterior near the root of the iris in either a clockwise or a counterclockwise direction to release PAS under direct view with the OE (Figure 1B). Both the main incision and a second incision were used to ensure all PAS areas were released. Complete synechialysis was confirmed under the direct view with the OE at the end of the procedure. Using an irrigation and aspiration handpiece from the phaco machine, balanced salt solution replaced the viscoelastic agent. The incision was closed by hydration or sutured with 10-0 nylon if necessary.

Patients used Pranoprofen eye drops (Senju Pharmaceutical Co., Ltd., Japan) and Levofloxacin eye drops (Santen, Japan) four times a day and 0.5% pilocarpine eyedrops (Bausch & Lomb, America) two times a day for four weeks after the surgery. Patients also used 1% prednisolone acetate eye drops (Allergan Pharmaceuticals, Ireland) four times a day for the first week after the surgery, and then reduced by one drop per week for a total of four weeks.

Success criteria Based on the AGIS study, we defined surgical success as follows: (1) Standard A: IOP<14mmHg using none or one type of IOP-lowering drug; (2) Standard B: IOP <18mmHg using none or one type of IOP-lowering drug.17 Statistical analysis All statistical analyses were performed using SPSS 20.0 statistical software. All data were represented by mean ± standard deviation (SD). The paired t-test was used to evaluate the differences in the extent of PAS, number of IOP lowering drugs, mean deviation , IOP and BCVA. A Spearman rank correlation coefficient was calculated to evaluate the correlation between the two groups of data.18 Statistical significance was set with a P-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

a diagnosis of PACG according to the International Society of Geographical & Epidemiological Ophthalmology (ISGEO) diagnostic criteria,[14] visual field score ≥18 calculated (as per the method used in the Advanced Glaucoma Intervention Study [AGIS]),[15] treatment with IOP-lowering drugs for more than 3 months, and mild to moderate cataract.

Exclusion Criteria:

secondary angle-closure glaucoma and previous history of surgery, except laser peripheral iridotomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The extent of peripheral anterior synechiae (PAS) | Change from Baseline PAS at 12 months
  observed the the extent of PAS before and after surgery
number of intraocular pressure (IOP) lowering drugs | Change from Baseline IOP lowering drugs at 12 months
  observed the the number of IOP lowering drugs before and after surgery
IOP | Change from Baseline IOP at 12 months
  IOP before and after surgery
best corrected visual acuity | Change from Baseline best corrected visual acuity at 12 months
  best corrected visual acuity before and after surgery
visual field | Change from Baseline MD of visual field at 12 months
  Mean defect（MD）of visual field before and after surgery